CLINICAL TRIAL: NCT00908869
Title: Combination of Continuous Low Doses of Vinorelbine, Cyclophosphamide and Interferon Alpha 2b for Antiangiogenic/Antivascular Effect in Adult Advanced Neoplasm
Brief Title: Combination of Continuous Low Doses of Vinorelbine, Cyclophosphamide and Interferon Alpha 2b (" Metronomic Chemotherapy ") for Antiangiogenic and Antivascular Effect. Trial With Pharmacodynamic Study in Adult Advanced Neoplasm
Acronym: METRO1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: METRO1/IPC2005-001
Record Dates: First submitted 2009-05-25; First posted 2009-05-27 (Estimated); Last update posted 2012-01-30 (Estimated); Status verified 2012-01

CONDITIONS: Advanced Neoplasm
Keywords: advanced neoplasm; adult advanced neoplasm
MeSH Terms: interventions — Vinorelbine; Cyclophosphamide; Interferon alpha-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Vinorelbine, Cyclophosphamide and Interferon alpha 2b — Level 1: Oral Vinorelbine (Navelbine®)20mg x 2/week; oral Cyclophosphamide (Endoxan®) 50mg/day; SC interferon alpha 2b (Introna®) 0.9 million IU x 3/week.
  Level 2: Oral Vinorelbine (Navelbine®)20mg x 3/week; oral Cyclophosphamide (Endoxan®) 50mg/day;SC interferon alpha 2b (Introna®) 0.9 million IU x 3/week.
  Level 3: Oral Vinorelbine (Navelbine®)20mg x 2/week; oral Cyclophosphamide (Endoxan®) 50mg/day; SC interferon alpha 2b (Introna®) 0.9 million IU x 5/week.
  Level -1 (in case of toxicity at level 1): Oral Vinorelbine (Navelbine®)20mg x 2/week; oral Cyclophosphamide (Endoxan®) 50mg/every 2 days; SC interferon alpha 2b (Introna®) 0.9 million IU x 3/week .

SUMMARY:
Purpose:

This phase I trial estimates the antiangiogenic and antivascular effect of 4 different levels of continuous low doses of the combination of Vinorelbine, Cyclophosphamide and Interferon alpha 2b (" metronomic chemotherapy ")in adult advanced neoplasm.

This study is non randomized, monocentric, and with a pharmacodynamic part.

Primary objective:

Estimation of the toxicity of the combination of continuous low doses of Vinorelbine, Cyclophosphamide and Interferon alpha 2b.

Secondary objectives:

Estimation of the antiangiogenic and/or antivascular effect (VEGF measurement) in radiography (DEC-MRI), biology and immunohistochemistry of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* patients aged from 18 and older,
* with metastatic or advanced solid tumor who received all standard treatments,
* who ended their chemotherapy or radiotherapy treatment within 4 weeks (6 weeks for mitocyne)prior entry in the study.
* All patients are included after being given written informed consent.

Exclusion Criteria:

* patients with stable disease,
* history or presence of another cancer,
* contraindication to administer the treatment,
* contraindication to perform MRI,
* pregnancy or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-05; Primary Completion 2010-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Estimation of the toxicity of the combination of continuous low doses of Vinorelbine, Cyclophosphamide and Interferon alpha 2b. | 6 weeks

SECONDARY OUTCOMES:
Estimation of the antiangiogenic and/or antivascular effect (VEGF measurement) in radiography (DEC-MRI), biology and immunohistochemistry of the treatment. | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Anthony GONCALVES, MD, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- Institut Paoli-Calmettes, Marseille, France

REFERENCES:
- See also: official site of the sponsor — http://www.institutpaolicalmettes.fr/